CLINICAL TRIAL: NCT07077876
Title: Surgical and Obstetric Outcomes in Patients With Endometrial Adenocarcinoma and Atypical Endometrial Hyperplasia Undergoing Conservative Treatment
Brief Title: Surgical and Obstetric Outcomes in Endometrial Adenocarcinoma and Atypical Endometrial Hyperplasia With Conservative Treatment
Acronym: CHOICE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Catena Ursula, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7309
Record Dates: First submitted 2025-06-26; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Hyperplasia; Fertility Preservation; Conservative Treatment Therapy
Keywords: Endometrial Cancer; Atypical Endometrial Hyperplasia; Fertility-Sparing Treatment; Hysteroscopy; Progestin Therapy; Reproductive Outcomes
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conservatively Treated Patients: Conservatively Treated Patients with Endometrial Cancer and Atypical Endometrial Hyperplasia
  Interventions: Procedure: Hysteroscopic Resection and Hormonal Therapy

INTERVENTIONS:
Procedure: Hysteroscopic Resection and Hormonal Therapy — Patients underwent hysteroscopic resection of atypical endometrial hyperplasia (AEH) or grade 1-2 endometrial adenocarcinoma (EAC) using a 15 Fr mini-resectoscope. Depending on the case, the procedure included visual D&C or a combined technique. At the end of the procedure, a 52 mg levonorgestrel-releasing intrauterine device (LNG-IUD) was inserted. In patients with EAC G2 or poor prognostic markers (e.g., MMR deficiency), oral progestin therapy with Megestrol Acetate (160 mg daily) was added. Follow-up included hysteroscopic endometrial biopsy at 3, 6, and 12 months to assess response.

SUMMARY:
This observational study aims to evaluate the obstetric and oncological outcomes of patients diagnosed with endometrial adenocarcinoma (EAC) or atypical endometrial hyperplasia (AEH) who underwent conservative treatment at the CLASS Hysteroscopy Center of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome. Eligible patients include women who received hysteroscopic surgery and hormonal therapy either to preserve fertility or due to medical contraindications to standard radical surgery. Follow-up lasts 12 months.

DETAILED DESCRIPTION:
This is a monocentric cohort study conducted at the CLASS Hysteroscopy Center of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome. It includes women diagnosed with endometrial adenocarcinoma (EAC) or atypical endometrial hyperplasia (AEH) who underwent conservative treatment using standardized hysteroscopic techniques performed by a single surgeon. The intervention consists of hysteroscopic lesion resection, insertion of a 52 mg levonorgestrel-releasing IUD, and in selected cases oral progestin therapy with Megestrol Acetate. The study includes both women desiring fertility preservation and patients medically unfit for radical surgery. Follow-up includes hysteroscopic biopsies at 3, 6, and 12 months. The primary objective is to assess obstetric outcomes, with secondary endpoints including oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older.
* Histological diagnosis of endometrial adenocarcinoma (EAC) or atypical endometrial hyperplasia (AEH).
* Patients who underwent conservative treatment with hysteroscopic resection at the CLASS Hysteroscopy Center, performed by a single experienced surgeon (U.C.).
* Patients treated conservatively due to medical contraindications to radical surgery (e.g., severe comorbidities).
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Patients with other known causes of infertility.
* Patients with non-endometrioid histological subtypes of endometrial adenocarcinoma.
* Patients under 18 years of age.
* Patients who did not provide informed consent for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with early-stage endometrial adenocarcinoma (EAC) or atypical endometrial hyperplasia (AEH) who underwent conservative hysteroscopic treatment at the CLASS Hysteroscopy Center of Fondazione Policlinico Universitario A. Gemelli IRCCS, either for fertility preservation or due to contraindications to radical surgery. All procedures were performed by a single experienced surgeon.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | Within 12 months from histologically confirmed complete response
  Proportion of participants who achieve a clinical pregnancy (intrauterine gestational sac with fetal heartbeat) after conservative treatment.
Miscarriage Rate | Within 12 months from histologically confirmed complete response
  Proportion of pregnancies that end in miscarriage (pregnancy loss < 20 weeks' gestation) among women who became pregnant after treatment.
Live Birth Rate | Within 12 months from histologically confirmed complete response
  Proportion of pregnancies resulting in at least one live-born infant after treatment.

SECONDARY OUTCOMES:
Disease-Free Interval | Up to 12 months after treatment
  Evaluation of time without disease recurrence from date of conservative treatment for EAC or AEH.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Catena, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catena U, Mirandola M, Capomacchia FM, Fanfani F, Scambia G. A new surgical approach for fertility-sparing management of diffuse endometrial G2 endometrioid adenocarcinoma: a step-by-step technique. Facts Views Vis Obgyn. 2023 Mar;15(1):79-81. doi: 10.52054/FVVO.15.1.058. PMID 37010338
- [Background] Morice P, Leary A, Creutzberg C, Abu-Rustum N, Darai E. Endometrial cancer. Lancet. 2016 Mar 12;387(10023):1094-1108. doi: 10.1016/S0140-6736(15)00130-0. Epub 2015 Sep 6. PMID 26354523
- [Background] Jeon YT, Park IA, Kim YB, Kim JW, Park NH, Kang SB, Lee HP, Song YS. Steroid receptor expressions in endometrial cancer: clinical significance and epidemiological implication. Cancer Lett. 2006 Aug 8;239(2):198-204. doi: 10.1016/j.canlet.2005.08.001. Epub 2005 Sep 15. PMID 16168561
- [Background] Di Spiezio Sardo A, De Angelis MC, Della Corte L, Carugno J, Zizolfi B, Guadagno E, Gencarelli A, Cecchi E, Simoncini T, Bifulco G, Zullo F, Insabato L. Should endometrial biopsy under direct hysteroscopic visualization using the grasp technique become the new gold standard for the preoperative evaluation of the patient with endometrial cancer? Gynecol Oncol. 2020 Aug;158(2):347-353. doi: 10.1016/j.ygyno.2020.05.012. Epub 2020 May 25. PMID 32467056
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338